CLINICAL TRIAL: NCT00309166
Title: An Observer-blind, Randomized, Controlled Study to Assess the Immunogenicity and Safety of GlaxoSmithKline Biologicals' HPV Vaccine Administered Intramuscularly According to a 0, 1, 6 Month Schedule in Healthy Male Subjects Aged 10-18 Years
Brief Title: Evaluation of the Immunogenicity and Safety of GlaxoSmithKline Biologicals' HPV Vaccine in Young Males.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 580299/011
Record Dates: First submitted 2006-03-28; First posted 2006-03-31 (Estimated); Results first posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-02

CONDITIONS: Infections, Papillomavirus
MeSH Terms: conditions — Papillomavirus Infections | interventions — human papillomavirus vaccine, L1 type 16, 18; Papillomavirus Vaccines

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Cervarix Group (Experimental): Healthy male subjects between and including 10 to 18 years of age at the time of the first vaccination, who were administered 3 doses of Cervarix™ (HPV-16/18 L1 VLP AS04) vaccine, intramuscularly into the deltoid region of the non-dominant arm, according to a 0, 1 and 6-month schedule. The subjects were followed up for 7 months after the first dose and an additional telephone contact was foreseen at Month 12.
  Interventions: Biological: Cervarix vaccine
- Engerix-B Group (Active Comparator): Healthy male subjects between and including 10 to 18 years of age at the time of the first vaccination, who were administered 3 doses of Engerix-B™ (HBV) vaccine, intramuscularly into the deltoid region of the non-dominant arm, according to a 0, 1 and 6-month schedule. The subjects were followed up for 7 months after the first dose and an additional telephone contact was foreseen at Month 12.
  Interventions: Biological: Engerix-B vaccine

INTERVENTIONS:
Biological: Cervarix vaccine — All subjects received an intramuscular injection into the deltoid of the non-dominant arm according to a 0, 1 and 6-month schedule.
  Other Names: HPV vaccine
  Arms: Cervarix Group
Biological: Engerix-B vaccine — All subjects received an intramuscular injection into the deltoid of the non-dominant arm according to a 0, 1 and 6-month schedule
  Other Names: HBV vaccine
  Arms: Engerix-B Group

SUMMARY:
The main aim of this vaccine is to prevent cervical cancer in women. However, it could also be relevant to vaccinate selected groups of males. Therefore, this study is designed to evaluate the safety and immunogenicity of the HPV vaccine in pre-teen and adolescent male subjects aged 10-18 years.

ELIGIBILITY:
Inclusion criteria:

* A male between, and including, 10 and 18 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject prior to enrolment
* For subjects below the legal age of consent, a written informed consent must be obtained from the subject's parent/guardian. In addition, a written informed assent must be obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Exclusion criteria:

* Previous vaccination against Human Papillomavirus (HPV).
* Previous vaccination against Hepatitis B, known clinical history of Hepatitis B infection.
* Cancer or autoimmune disease under treatment.

Ages: 10 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 270 (Actual)
Dates: Start 2006-04-05 (Actual); Primary Completion 2007-06-01 (Actual); Study Completion 2007-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Finland (5):
  - GSK Investigational Site, Kotka
  - GSK Investigational Site, Kouvola
  - GSK Investigational Site, Mikkeli
  - GSK Investigational Site, Rauma
  - GSK Investigational Site, Tampere

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Petaja T, Keranen H, Karppa T, Kawa A, Lantela S, Siitari-Mattila M, Levanen H, Tocklin T, Godeaux O, Lehtinen M, Dubin G. Immunogenicity and safety of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine in healthy boys aged 10-18 years. J Adolesc Health. 2009 Jan;44(1):33-40. doi: 10.1016/j.jadohealth.2008.10.002. PMID 19101456
- [Background] Verstraeten T, Descamps D, David MP, Zahaf T, Hardt K, Izurieta P, Dubin G, Breuer T. Analysis of adverse events of potential autoimmune aetiology in a large integrated safety database of AS04 adjuvanted vaccines. Vaccine. 2008 Dec 2;26(51):6630-8. doi: 10.1016/j.vaccine.2008.09.049. PMID 18845199
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 580299/011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 580299/011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 580299/011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 580299/011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 580299/011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 580299/011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Period: Overall Study
Arm/Group | Cervarix Group | Engerix-B Group
Started | 181 | 89
Completed | 176 | 86
Not Completed | 5 | 3
Not completed — Adverse event, non-fatal | 1 | 0
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Group | Engerix-B Group | Total
Number analyzed (Participants) | 181 | 89 | 270
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.4 (2.14) | 14.4 (2.02) | 14.4 (2.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 181 | 89 | 270
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African heritage/African American | 1 | 0 | 1
  Geographic ancestry: Asian-Central/South Asian heritage | 1 | 0 | 1
  Geographic ancestry: White-Arabic/North African heritage | 1 | 0 | 1
  Geographic ancestry: White-Caucasian/European heritage | 177 | 88 | 265
  Geographic ancestry: Not specified | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects for Anti-HPV-16 and Anti-HPV-18
Description: Seroconversion was defined as the appearance of anti-HPV-16 and/or anti-HPV-18 antibodies [anti-HPV-16 titers greater than or equal to (≥) 8 enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL) and anti-HPV-18 titres ≥7 EL.U/mL] in the serum of subjects seronegative before vaccination.
Time Frame: At Month 7
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Engerix-B Group
Number analyzed (Participants) | 163 | 86
Participants
  HPV-16: number analyzed (Participants) | 163 | 83
  HPV-16 | 163 | 1
  HPV-18: number analyzed (Participants) | 150 | 86
  HPV-18 | 150 | 2

2. Primary Outcome: Antibody Titers Against HPV-16 (Anti-HPV-16) and HPV-18 (Anti-HPV-18)
Description: Titers were presented as geometric mean titers (GMT).
Time Frame: At Month 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Engerix-B Group
Number analyzed (Participants) | 171 | 86
EL.U/mL
  HPV-16 | 22564.8 [19800.3 to 25715.4] | 4.2 [4.0 to 4.5]
  HPV-18: number analyzed (Participants) | 170 | 86
  HPV-18 | 8460.3 [7306.1 to 9796.8] | 3.6 [3.4 to 3.8]

3. Secondary Outcome: Number of Seroconverted Subjects for Anti-HPV-16 and Anti-HPV-18
Description: Seroconversion was defined as the appearance of anti-HPV-16 and/or anti-HPV-18 antibodies (anti-HPV-16 titres ≥ 8 EL.U/mL and anti-HPV-18 titres ≥ 7 EL.U/mL) in the serum of subjects seronegative before vaccination.
Time Frame: At Month 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Engerix-B Group
Number analyzed (Participants) | 165 | 86
Participants
  HPV-16: number analyzed (Participants) | 165 | 83
  HPV-16 | 165 | 0
  HPV-18: number analyzed (Participants) | 152 | 86
  HPV-18 | 152 | 4

4. Secondary Outcome: Antibody Titers Against HPV-16 (Anti-HPV-16) and HPV-18 (Anti-HPV-18)
Description: Titers were presented as GMTs.
Time Frame: At Month 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Engerix-B Group
Number analyzed (Participants) | 173 | 86
EL.U/mL
  HPV-16 | 5254.5 [4704.9 to 5868.2] | 4.1 [4 to 4.3]
  HPV-18: number analyzed (Participants) | 172 | 86
  HPV-18 | 3696.9 [3275.9 to 4172.1] | 3.7 [3.5 to 3.8]

5. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = any solicited local symptom irrespective of intensity grade; Grade 3 pain = pain that prevented normal activity; Grade 3 redness/swelling = redness/swelling spreading beyond (>) 50 mm.
Time Frame: Within 7 days (Days 0-6) after each dose and across doses, up to 7 months
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available and who had filled in the symptom sheet.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Engerix-B Group
Number analyzed (Participants) | 180 | 88
Participants
  Pain, Dose 1 | 149 | 25
  Grade 3 Pain, Dose 1 | 1 | 0
  Redness, Dose 1 | 24 | 12
  Grade 3 Redness, Dose 1 | 0 | 0
  Swelling, Dose 1 | 7 | 3
  Grade 3 Swelling, Dose 1 | 0 | 0
  Pain, Dose 2: number analyzed (Participants) | 172 | 86
  Pain, Dose 2 | 114 | 16
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 172 | 86
  Grade 3 Pain, Dose 2 | 2 | 0
  Redness, Dose 2: number analyzed (Participants) | 172 | 86
  Redness, Dose 2 | 30 | 8
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 172 | 86
  Grade 3 Redness, Dose 2 | 0 | 0
  Swelling, Dose 2: number analyzed (Participants) | 172 | 86
  Swelling, Dose 2 | 20 | 2
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 172 | 86
  Grade 3 Swelling, Dose 2 | 0 | 1
  Pain, Dose 3: number analyzed (Participants) | 171 | 85
  Pain, Dose 3 | 115 | 16
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 171 | 85
  Grade 3 Pain, Dose 3 | 7 | 0
  Redness, Dose 3: number analyzed (Participants) | 171 | 85
  Redness, Dose 3 | 33 | 9
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 171 | 85
  Grade 3 Redness, Dose 3 | 0 | 0
  Swelling, Dose 3: number analyzed (Participants) | 171 | 85
  Swelling, Dose 3 | 29 | 3
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 171 | 85
  Grade 3 Swelling, Dose 3 | 2 | 0
  Pain, Across doses | 159 | 39
  Grade 3 Pain, Across doses | 8 | 0
  Redness, Across doses | 51 | 15
  Grade 3 Redness, Across doses | 0 | 0
  Swelling, Across doses | 36 | 7
  Grade 3 Swelling, Across doses | 2 | 1

6. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed were arthralgia, fatigue, fever (defined as axillary temperature ≥37.5 °C), gastrointestinal, headache, myalgia, rash and urticaria. Any = any solicited general symptom irrespective of intensity grade or relationship to vaccination; Grade 3 = symptom that prevented normal activity; Grade 3 fever = temperature > 39.0 °C; Related = symptoms considered by the investigator to have a causal relationship to vaccination.
Time Frame: Within 7 days (Days 0-6) after each dose and across doses, up to 7 months
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available and who had filled in the symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Engerix-B Group
Number analyzed (Participants) | 180 | 88
Participants
  Arthralgia, Dose 1 | 17 | 7
  Grade 3 Athralgia, Dose 1 | 0 | 0
  Related Athralgia, Dose 1 | 10 | 3
  Fatigue, Dose 1 | 51 | 32
  Grade 3 Fatigue, Dose 1 | 1 | 0
  Related Fatigue, Dose 1 | 26 | 18
  Fever (axillary), Dose 1 | 24 | 11
  Grade 3 Fever, Dose 1 | 0 | 0
  Related Fever, Dose 1 | 1 | 1
  Gastrointestinal, Dose 1 | 33 | 10
  Grade 3 Gastrointestinal, Dose 1 | 2 | 0
  Related Gastrointestinal, Dose 1 | 15 | 5
  Headache, Dose 1 | 51 | 21
  Grade 3 Headache, Dose 1 | 0 | 0
  Related Headache, Dose 1 | 24 | 7
  Myalgia, Dose 1 | 67 | 16
  Grade 3 Mylagia, Dose 1 | 1 | 0
  Related Mylagia, Dose 1 | 45 | 7
  Rash, Dose 1 | 8 | 1
  Grade 3 Rash, Dose 1 | 0 | 0
  Related Rash, Dose 1 | 2 | 1
  Urticaria, Dose 1 | 3 | 0
  Grade 3 Urticaria, Dose 1 | 0 | 0
  Related Urticaria, Dose 1 | 1 | 0
  Arthralgia, Dose 2: number analyzed (Participants) | 173 | 86
  Arthralgia, Dose 2 | 6 | 3
  Grade 3 Arthralgia, Dose 2: number analyzed (Participants) | 173 | 86
  Grade 3 Arthralgia, Dose 2 | 0 | 1
  Related Arthralgia, Dose 2: number analyzed (Participants) | 173 | 86
  Related Arthralgia, Dose 2 | 3 | 0
  Fatigue, Dose 2: number analyzed (Participants) | 173 | 86
  Fatigue, Dose 2 | 35 | 14
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 173 | 86
  Grade 3 Fatigue, Dose 2 | 1 | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 173 | 86
  Related Fatigue, Dose 2 | 21 | 9
  Fever (axillary), Dose 2: number analyzed (Participants) | 173 | 86
  Fever (axillary), Dose 2 | 14 | 6
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 173 | 86
  Grade 3 Fever, Dose 2 | 0 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 173 | 86
  Related Fever, Dose 2 | 1 | 0
  Gastrointestinal, Dose 2: number analyzed (Participants) | 173 | 86
  Gastrointestinal, Dose 2 | 18 | 4
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 173 | 86
  Grade 3 Gastrointestinal, Dose 2 | 1 | 1
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 173 | 86
  Related Gastrointestinal, Dose 2 | 7 | 0
  Headache, Dose 2: number analyzed (Participants) | 173 | 86
  Headache, Dose 2 | 30 | 13
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 173 | 86
  Grade 3 Headache, Dose 2 | 2 | 1
  Related Headache, Dose 2: number analyzed (Participants) | 173 | 86
  Related Headache, Dose 2 | 14 | 7
  Myalgia, Dose 2: number analyzed (Participants) | 173 | 86
  Myalgia, Dose 2 | 35 | 8
  Grade 3 Maylagia, Dose 2: number analyzed (Participants) | 173 | 86
  Grade 3 Maylagia, Dose 2 | 1 | 0
  Related Maylagia, Dose 2: number analyzed (Participants) | 173 | 86
  Related Maylagia, Dose 2 | 27 | 7
  Rash, Dose 2: number analyzed (Participants) | 173 | 86
  Rash, Dose 2 | 8 | 2
  Grade 3 Rash, Dose 2: number analyzed (Participants) | 173 | 86
  Grade 3 Rash, Dose 2 | 0 | 0
  Related Rash, Dose 2: number analyzed (Participants) | 173 | 86
  Related Rash, Dose 2 | 3 | 0
  Urticaria, Dose 2: number analyzed (Participants) | 173 | 86
  Urticaria, Dose 2 | 1 | 2
  Grade 3 Urticaria, Dose 2: number analyzed (Participants) | 173 | 86
  Grade 3 Urticaria, Dose 2 | 0 | 0
  Related Urticaria, Dose 2: number analyzed (Participants) | 173 | 86
  Related Urticaria, Dose 2 | 0 | 0
  Arthralgia, Dose 3: number analyzed (Participants) | 170 | 85
  Arthralgia, Dose 3 | 12 | 3
  Grade 3 Arthralgia, Dose 3: number analyzed (Participants) | 170 | 85
  Grade 3 Arthralgia, Dose 3 | 0 | 0
  Related Arthtralgia, Dose 3: number analyzed (Participants) | 170 | 85
  Related Arthtralgia, Dose 3 | 12 | 3
  Fatigue, Dose 3: number analyzed (Participants) | 170 | 85
  Fatigue, Dose 3 | 44 | 15
  Grade 3 Fatigue, Dose 3: number analyzed (Participants) | 170 | 85
  Grade 3 Fatigue, Dose 3 | 2 | 0
  Related Fatigue, Dose 3: number analyzed (Participants) | 170 | 85
  Related Fatigue, Dose 3 | 30 | 11
  Fever (axillary), Dose 3: number analyzed (Participants) | 170 | 85
  Fever (axillary), Dose 3 | 14 | 4
  Grade 3 Fever, Dose 3: number analyzed (Participants) | 170 | 85
  Grade 3 Fever, Dose 3 | 0 | 0
  Related Fever, Dose 3: number analyzed (Participants) | 170 | 85
  Related Fever, Dose 3 | 1 | 0
  Gastrointestinal, Dose 3: number analyzed (Participants) | 170 | 85
  Gastrointestinal, Dose 3 | 10 | 5
  Grade 3 Gastrointestinal, Dose 3: number analyzed (Participants) | 170 | 85
  Grade 3 Gastrointestinal, Dose 3 | 1 | 0
  Related Gastrointestinal, Dose 3: number analyzed (Participants) | 170 | 85
  Related Gastrointestinal, Dose 3 | 8 | 4
  Headache, Dose 3: number analyzed (Participants) | 170 | 85
  Headache, Dose 3 | 30 | 11
  Grade 3 Headache, Dose 3: number analyzed (Participants) | 170 | 85
  Grade 3 Headache, Dose 3 | 3 | 0
  Related Headache, Dose 3: number analyzed (Participants) | 170 | 85
  Related Headache, Dose 3 | 17 | 8
  Myalgia, Dose 3: number analyzed (Participants) | 170 | 85
  Myalgia, Dose 3 | 39 | 8
  Grade 3 Mylagia, Dose 3: number analyzed (Participants) | 170 | 85
  Grade 3 Mylagia, Dose 3 | 1 | 0
  Related Mylagia, Dose 3: number analyzed (Participants) | 170 | 85
  Related Mylagia, Dose 3 | 35 | 6
  Rash, Dose 3: number analyzed (Participants) | 170 | 85
  Rash, Dose 3 | 3 | 2
  Grade 3 Rash, Dose 3: number analyzed (Participants) | 170 | 85
  Grade 3 Rash, Dose 3 | 0 | 0
  Related Rash, Dose 3: number analyzed (Participants) | 170 | 85
  Related Rash, Dose 3 | 1 | 0
  Urticaria, Dose 3: number analyzed (Participants) | 170 | 85
  Urticaria, Dose 3 | 0 | 0
  Grade 3 Urticaria, Dose 3: number analyzed (Participants) | 170 | 85
  Grade 3 Urticaria, Dose 3 | 0 | 0
  Related Urticaria, Dose 3: number analyzed (Participants) | 170 | 85
  Related Urticaria, Dose 3 | 0 | 0
  Arthralgia, Across doses | 29 | 10
  Grade 3 Arthralgia, Across doses | 0 | 1
  Related Arthralgia, Across doses | 22 | 5
  Fatigue, Across doses | 82 | 42
  Grade 3 Fatigue, Across doses | 4 | 0
  Related Fatigue, Across doses | 52 | 33
  Fever (axillary), Across doses | 35 | 17
  Grade 3 Fever, Across doses | 0 | 0
  Related Fever, Across doses | 3 | 1
  Gastrointestinal, Across doses | 40 | 14
  Grade 3 Gastrointestinal, Across doses | 4 | 1
  Related Gastrointestinal, Across doses | 19 | 7
  Headache, Across doses | 77 | 33
  Grade 3 Headache, Across doses | 5 | 1
  Related Headache, Across doses | 43 | 16
  Myalgia, Across doses | 88 | 23
  Grade 3 Mylagia, Across doses | 3 | 0
  Related Mylagia, Across doses | 70 | 14
  Rash, Across doses | 16 | 5
  Grade 3 Rash, Across doses | 0 | 0
  Related Rash, Across doses | 5 | 1
  Urticaria, Across doses | 4 | 2
  Grade 3 Urticaria, Across doses | 0 | 0
  Related Urticaria, Across doses | 1 | 0

7. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within 30 days (Day 0-29) after any vaccination, up to 7 months
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Engerix-B Group
Number analyzed (Participants) | 181 | 89
Participants
  Any AEs | 68 | 31
  Grade 3 AEs | 5 | 2
  Related AEs | 5 | 1

8. Secondary Outcome: Number of Subjects With New Onset of Chronic Diseases (NOCDs) and Other Medically Significant Conditions
Description: NOCDs include asthma, Chron's disease, dermatitis atopic. MSCs include AEs prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections and injury.
Time Frame: Throughout the active phase of the study (up to Month 7) and the extended safety follow-up (from Month 7 up to Month 12)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available up to Month 7 and on the Extended Safety Follow-Up (ESFU) Total Vaccinated cohort, which included all vaccinated subjects that could be contacted by telephone for the Safety follow-up at Month 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Engerix-B Group
Number analyzed (Participants) | 181 | 89
Participants
  NOCDs, Month 7 | 2 | 1
  MSCs, Month 7 | 22 | 10
  NOCDs, Month 7 to Month 12: number analyzed (Participants) | 175 | 86
  NOCDs, Month 7 to Month 12 | 0 | 0
  MSCs, Month 7 to Month 12: number analyzed (Participants) | 175 | 86
  MSCs, Month 7 to Month 12 | 1 | 2

9. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Engerix-B Group
Number analyzed (Participants) | 181 | 89
Participants
  SAEs, Month 7 | 2 | 0
  SAEs, Month 12: number analyzed (Participants) | 175 | 86
  SAEs, Month 12 | 1 | 1

10. Secondary Outcome: Number of Subjects With Clinically Relevant Abnormalities in Biochemical and Haematological Parameters
Description: The occurence of clinically relevant abnormalities was assessed in the following biochemical and haematological parameters: alanine aminotransferase [ALT], basophils [BAS], creatinine [CREA], eosinophils [EOS] and hematocrit [Hem]. Levels of haematological/biochemical parameters assessed in terms of normal, below and above laboratory values were - normal, below, above and missing.
Time Frame: At Month 2 and Month 7, post-vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Engerix-B Group
Number analyzed (Participants) | 172 | 86
Participants
  ALT Normal, Month 2, Normal | 166 | 79
  ALT Normal, Month 2, Below | 3 | 0
  ALT Normal, Month 2, Above | 3 | 2
  ALT Normal, Month 2, Missing | 0 | 5
  ALT Normal, Month 7, Normal: number analyzed (Participants) | 171 | 84
  ALT Normal, Month 7, Normal | 165 | 81
  ALT Normal, Month 7, Below: number analyzed (Participants) | 171 | 84
  ALT Normal, Month 7, Below | 1 | 0
  ALT Normal, Month 7, Above: number analyzed (Participants) | 171 | 84
  ALT Normal, Month 7, Above | 5 | 3
  ALT Below, Month 2, Normal: number analyzed (Participants) | 1 | 0
  ALT Below, Month 2, Normal | 0 | 0
  ALT Below, Month 2, Below: number analyzed (Participants) | 1 | 0
  ALT Below, Month 2, Below | 1 | 0
  ALT Below, Month 2, Above: number analyzed (Participants) | 1 | 0
  ALT Below, Month 2, Above | 0 | 0
  ALT Below, Month 7, Normal: number analyzed (Participants) | 1 | 0
  ALT Below, Month 7, Normal | 0 | 0
  ALT Below, Month 7, Below: number analyzed (Participants) | 1 | 0
  ALT Below, Month 7, Below | 1 | 0
  ALT Below, Month 7, Above: number analyzed (Participants) | 1 | 0
  ALT Below, Month 7, Above | 0 | 0
  ALT Above, Month 2, Normal: number analyzed (Participants) | 4 | 1
  ALT Above, Month 2, Normal | 2 | 0
  ALT Above, Month 2, Below: number analyzed (Participants) | 4 | 1
  ALT Above, Month 2, Below | 0 | 0
  ALT Above, Month 2, Above: number analyzed (Participants) | 4 | 1
  ALT Above, Month 2, Above | 2 | 0
  ALT Above, Month 2, Missing: number analyzed (Participants) | 4 | 1
  ALT Above, Month 2, Missing | 0 | 1
  ALT Above, Month 7, Normal: number analyzed (Participants) | 3 | 1
  ALT Above, Month 7, Normal | 2 | 0
  ALT Above, Month 7, Below: number analyzed (Participants) | 3 | 1
  ALT Above, Month 7, Below | 0 | 0
  ALT Above, Month 7, Above: number analyzed (Participants) | 3 | 1
  ALT Above, Month 7, Above | 1 | 1
  BAS Normal, Month 2, Normal: number analyzed (Participants) | 146 | 76
  BAS Normal, Month 2, Normal | 140 | 65
  BAS Normal, Month 2, Below: number analyzed (Participants) | 146 | 76
  BAS Normal, Month 2, Below | 0 | 0
  BAS Normal, Month 2, Above: number analyzed (Participants) | 146 | 76
  BAS Normal, Month 2, Above | 3 | 3
  BAS Normal, Month 2, Missing: number analyzed (Participants) | 146 | 76
  BAS Normal, Month 2, Missing | 3 | 8
  BAS Normal, Month 7, Normal: number analyzed (Participants) | 145 | 74
  BAS Normal, Month 7, Normal | 134 | 66
  BAS Normal, Month 7, Below: number analyzed (Participants) | 145 | 74
  BAS Normal, Month 7, Below | 0 | 0
  BAS Normal, Month 7, Above: number analyzed (Participants) | 145 | 74
  BAS Normal, Month 7, Above | 11 | 8
  BAS Above, Month 2, Normal: number analyzed (Participants) | 18 | 6
  BAS Above, Month 2, Normal | 12 | 5
  BAS Above, Month 2, Below: number analyzed (Participants) | 18 | 6
  BAS Above, Month 2, Below | 0 | 0
  BAS Above, Month 2, Above: number analyzed (Participants) | 18 | 6
  BAS Above, Month 2, Above | 6 | 1
  BAS Above, Month 7, Normal: number analyzed (Participants) | 18 | 6
  BAS Above, Month 7, Normal | 14 | 4
  BAS Above, Month 7, Below: number analyzed (Participants) | 18 | 6
  BAS Above, Month 7, Below | 0 | 0
  BAS Above, Month 7, Above: number analyzed (Participants) | 18 | 6
  BAS Above, Month 7, Above | 4 | 2
  EOS Normal, Month 2, Normal: number analyzed (Participants) | 125 | 68
  EOS Normal, Month 2, Normal | 102 | 48
  EOS Normal, Month 2, Below: number analyzed (Participants) | 125 | 68
  EOS Normal, Month 2, Below | 4 | 2
  EOS Normal, Month 2, Above: number analyzed (Participants) | 125 | 68
  EOS Normal, Month 2, Above | 17 | 10
  EOS Normal, Month 2, Missing: number analyzed (Participants) | 125 | 68
  EOS Normal, Month 2, Missing | 2 | 8
  EOS Normal, Month 7, Normal: number analyzed (Participants) | 125 | 67
  EOS Normal, Month 7, Normal | 108 | 54
  EOS Normal, Month 7, Below: number analyzed (Participants) | 125 | 67
  EOS Normal, Month 7, Below | 8 | 4
  EOS Normal, Month 7, Above: number analyzed (Participants) | 125 | 67
  EOS Normal, Month 7, Above | 9 | 9
  EOS Below, Month 2, Normal: number analyzed (Participants) | 4 | 3
  EOS Below, Month 2, Normal | 4 | 2
  EOS Below, Month 2, Below: number analyzed (Participants) | 4 | 3
  EOS Below, Month 2, Below | 0 | 1
  EOS Below, Month 2, Above: number analyzed (Participants) | 4 | 3
  EOS Below, Month 2, Above | 0 | 0
  EOS Below, Month 7, Normal: number analyzed (Participants) | 4 | 2
  EOS Below, Month 7, Normal | 2 | 1
  EOS Below, Month 7, Below: number analyzed (Participants) | 4 | 2
  EOS Below, Month 7, Below | 2 | 1
  EOS Below, Month 7, Above: number analyzed (Participants) | 4 | 2
  EOS Below, Month 7, Above | 0 | 0
  EOS Above, Month 2, Normal: number analyzed (Participants) | 36 | 11
  EOS Above, Month 2, Normal | 6 | 5
  EOS Above, Month 2, Below: number analyzed (Participants) | 36 | 11
  EOS Above, Month 2, Below | 0 | 0
  EOS Above, Month 2, Above: number analyzed (Participants) | 36 | 11
  EOS Above, Month 2, Above | 30 | 6
  EOS Above, Month 7, Normal: number analyzed (Participants) | 35 | 11
  EOS Above, Month 7, Normal | 8 | 5
  EOS Above, Month 7, Below: number analyzed (Participants) | 35 | 11
  EOS Above, Month 7, Below | 0 | 0
  EOS Above, Month 7, Above: number analyzed (Participants) | 35 | 11
  EOS Above, Month 7, Above | 27 | 6
  CREA Normal, Month 2, Normal: number analyzed (Participants) | 163 | 82
  CREA Normal, Month 2, Normal | 158 | 76
  CREA Normal, Month 2, Below: number analyzed (Participants) | 163 | 82
  CREA Normal, Month 2, Below | 0 | 0
  CREA Normal, Month 2, Above: number analyzed (Participants) | 163 | 82
  CREA Normal, Month 2, Above | 5 | 0
  CREA Normal, Month 2, Missing: number analyzed (Participants) | 163 | 82
  CREA Normal, Month 2, Missing | 0 | 6
  CREA Normal, Month 7, Normal: number analyzed (Participants) | 161 | 80
  CREA Normal, Month 7, Normal | 159 | 79
  CREA Normal, Month 7, Below: number analyzed (Participants) | 161 | 80
  CREA Normal, Month 7, Below | 0 | 0
  CREA Normal, Month 7, Above: number analyzed (Participants) | 161 | 80
  CREA Normal, Month 7, Above | 2 | 1
  CREA Above, Month 2, Normal: number analyzed (Participants) | 13 | 5
  CREA Above, Month 2, Normal | 10 | 3
  CREA Above, Month 2, Below: number analyzed (Participants) | 13 | 5
  CREA Above, Month 2, Below | 0 | 0
  CREA Above, Month 2, Above: number analyzed (Participants) | 13 | 5
  CREA Above, Month 2, Above | 3 | 2
  CREA Above, Month 7, Normal: number analyzed (Participants) | 13 | 5
  CREA Above, Month 7, Normal | 10 | 5
  CREA Above, Month 7, Below: number analyzed (Participants) | 13 | 5
  CREA Above, Month 7, Below | 0 | 0
  CREA Above, Month 7, Above: number analyzed (Participants) | 13 | 5
  CREA Above, Month 7, Above | 3 | 0
  HEM Normal, Month 2, Normal: number analyzed (Participants) | 159 | 81
  HEM Normal, Month 2, Normal | 155 | 76
  HEM Normal, Month 2, Below: number analyzed (Participants) | 159 | 81
  HEM Normal, Month 2, Below | 2 | 0
  HEM Normal, Month 2, Above: number analyzed (Participants) | 159 | 81
  HEM Normal, Month 2, Above | 2 | 0
  HEM Normal, Month 2, Missing: number analyzed (Participants) | 159 | 81
  HEM Normal, Month 2, Missing | 0 | 5
  HEM Normal, Month 7, Normal: number analyzed (Participants) | 158 | 79
  HEM Normal, Month 7, Normal | 147 | 73
  HEM Normal, Month 7, Below: number analyzed (Participants) | 158 | 79
  HEM Normal, Month 7, Below | 9 | 6
  HEM Normal, Month 7, Above: number analyzed (Participants) | 158 | 79
  HEM Normal, Month 7, Above | 2 | 0
  HEM Below, Month 2, Normal: number analyzed (Participants) | 4 | 1
  HEM Below, Month 2, Normal | 3 | 1
  HEM Below, Month 2, Below: number analyzed (Participants) | 4 | 1
  HEM Below, Month 2, Below | 1 | 0
  HEM Below, Month 2, Above: number analyzed (Participants) | 4 | 1
  HEM Below, Month 2, Above | 0 | 0
  HEM Below, Month 7, Normal: number analyzed (Participants) | 4 | 1
  HEM Below, Month 7, Normal | 2 | 1
  HEM Below, Month 7, Below: number analyzed (Participants) | 4 | 1
  HEM Below, Month 7, Below | 2 | 0
  HEM Below, Month 7, Above: number analyzed (Participants) | 4 | 1
  HEM Below, Month 7, Above | 0 | 0
  HEM Above, Month 2, Normal: number analyzed (Participants) | 6 | 2
  HEM Above, Month 2, Normal | 3 | 0
  HEM Above, Month 2, Below: number analyzed (Participants) | 6 | 2
  HEM Above, Month 2, Below | 0 | 0
  HEM Above, Month 2, Above: number analyzed (Participants) | 6 | 2
  HEM Above, Month 2, Above | 3 | 1
  HEM Above, Month 2, Missing: number analyzed (Participants) | 6 | 2
  HEM Above, Month 2, Missing | 0 | 1
  HEM Above, Month 7, Normal: number analyzed (Participants) | 6 | 2
  HEM Above, Month 7, Normal | 6 | 1
  HEM Above, Month 7, Below: number analyzed (Participants) | 6 | 2
  HEM Above, Month 7, Below | 0 | 0
  HEM Above, Month 7, Above: number analyzed (Participants) | 6 | 2
  HEM Above, Month 7, Above | 0 | 1

11. Secondary Outcome: Number of Subjects With Clinically Relevant Abnormalities in Biochemical and Haematological Parameters
Description: The occurence of clinically relevant abnormalities was assessed in the following biochemical and haematological parameters: lymphocytes [LYM], monocytes [MON], neutrophils [NEU], platelets [PLA], red blood cells [RBC] and white blood cells [WBC]. Levels of haematological/biochemical parameters assessed in terms of normal, below and above laboratory values were - normal, below, above and missing.
Time Frame: At Month 2 and at Month 7, post-vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Engerix-B Group
Number analyzed (Participants) | 164 | 82
Participants
  LYM Normal, Month 2, Normal: number analyzed (Participants) | 142 | 71
  LYM Normal, Month 2, Normal | 117 | 56
  LYM Normal, Month 2, Below: number analyzed (Participants) | 142 | 71
  LYM Normal, Month 2, Below | 5 | 1
  LYM Normal, Month 2, Above: number analyzed (Participants) | 142 | 71
  LYM Normal, Month 2, Above | 18 | 6
  LYM Normal, Month 2, Missing: number analyzed (Participants) | 142 | 71
  LYM Normal, Month 2, Missing | 2 | 8
  LYM Normal, Month 7, Normal: number analyzed (Participants) | 142 | 69
  LYM Normal, Month 7, Normal | 126 | 63
  LYM Normal, Month 7, Below: number analyzed (Participants) | 142 | 69
  LYM Normal, Month 7, Below | 4 | 1
  LYM Normal, Month 7, Above: number analyzed (Participants) | 142 | 69
  LYM Normal, Month 7, Above | 12 | 5
  LYM Below, Month 2, Normal: number analyzed (Participants) | 3 | 1
  LYM Below, Month 2, Normal | 1 | 1
  LYM Below, Month 2, Below: number analyzed (Participants) | 3 | 1
  LYM Below, Month 2, Below | 2 | 0
  LYM Below, Month 2, Above: number analyzed (Participants) | 3 | 1
  LYM Below, Month 2, Above | 0 | 0
  LYM Below, Month 7, Normal: number analyzed (Participants) | 3 | 1
  LYM Below, Month 7, Normal | 2 | 1
  LYM Below, Month 7, Below: number analyzed (Participants) | 3 | 1
  LYM Below, Month 7, Below | 1 | 0
  LYM Below, Month 7, Above: number analyzed (Participants) | 3 | 1
  LYM Below, Month 7, Above | 0 | 0
  LYM Above, Month 2, Normal: number analyzed (Participants) | 20 | 10
  LYM Above, Month 2, Normal | 11 | 5
  LYM Above, Month 2, Below: number analyzed (Participants) | 20 | 10
  LYM Above, Month 2, Below | 1 | 0
  LYM Above, Month 2, Above: number analyzed (Participants) | 20 | 10
  LYM Above, Month 2, Above | 8 | 5
  LYM Above, Month 7, Normal: number analyzed (Participants) | 19 | 10
  LYM Above, Month 7, Normal | 11 | 8
  LYM Above, Month 7, Below: number analyzed (Participants) | 19 | 10
  LYM Above, Month 7, Below | 0 | 0
  LYM Above, Month 7, Above: number analyzed (Participants) | 19 | 10
  LYM Above, Month 7, Above | 8 | 2
  MON Normal, Month 2, Normal: number analyzed (Participants) | 108 | 50
  MON Normal, Month 2, Normal | 92 | 38
  MON Normal, Month 2, Below: number analyzed (Participants) | 108 | 50
  MON Normal, Month 2, Below | 0 | 0
  MON Normal, Month 2, Above: number analyzed (Participants) | 108 | 50
  MON Normal, Month 2, Above | 15 | 5
  MON Normal, Month 2, Missing: number analyzed (Participants) | 108 | 50
  MON Normal, Month 2, Missing | 1 | 7
  MON Normal, Month 7, Normal: number analyzed (Participants) | 108 | 48
  MON Normal, Month 7, Normal | 93 | 43
  MON Normal, Month 7, Below: number analyzed (Participants) | 108 | 48
  MON Normal, Month 7, Below | 0 | 1
  MON Normal, Month 7, Above: number analyzed (Participants) | 108 | 48
  MON Normal, Month 7, Above | 15 | 4
  MON Below, Month 2, Normal: number analyzed (Participants) | 1 | 3
  MON Below, Month 2, Normal | 1 | 3
  MON Below, Month 2, Below: number analyzed (Participants) | 1 | 3
  MON Below, Month 2, Below | 0 | 0
  MON Below, Month 2, Above: number analyzed (Participants) | 1 | 3
  MON Below, Month 2, Above | 0 | 0
  MON Below, Month 7, Normal: number analyzed (Participants) | 1 | 3
  MON Below, Month 7, Normal | 0 | 3
  MON Below, Month 7, Below: number analyzed (Participants) | 1 | 3
  MON Below, Month 7, Below | 1 | 0
  MON Below, Month 7, Above: number analyzed (Participants) | 1 | 3
  MON Below, Month 7, Above | 0 | 0
  MON Above, Month 2, Normal: number analyzed (Participants) | 56 | 29
  MON Above, Month 2, Normal | 7 | 8
  MON Above, Month 2, Below: number analyzed (Participants) | 56 | 29
  MON Above, Month 2, Below | 0 | 0
  MON Above, Month 2, Above: number analyzed (Participants) | 56 | 29
  MON Above, Month 2, Above | 48 | 20
  MON Above, Month 2, Missing: number analyzed (Participants) | 56 | 29
  MON Above, Month 2, Missing | 1 | 1
  MON Above, Month 7, Normal: number analyzed (Participants) | 55 | 29
  MON Above, Month 7, Normal | 13 | 7
  MON Above, Month 7, Below: number analyzed (Participants) | 55 | 29
  MON Above, Month 7, Below | 0 | 0
  MON Above, Month 7, Above: number analyzed (Participants) | 55 | 29
  MON Above, Month 7, Above | 42 | 22
  NEU Normal, Month 2, Normal: number analyzed (Participants) | 152 | 74
  NEU Normal, Month 2, Normal | 130 | 60
  NEU Normal, Month 2, Below: number analyzed (Participants) | 152 | 74
  NEU Normal, Month 2, Below | 20 | 6
  NEU Normal, Month 2, Above: number analyzed (Participants) | 152 | 74
  NEU Normal, Month 2, Above | 0 | 0
  NEU Normal, Month 2, Missing: number analyzed (Participants) | 152 | 74
  NEU Normal, Month 2, Missing | 2 | 8
  NEU Normal, Month 7, Normal: number analyzed (Participants) | 152 | 72
  NEU Normal, Month 7, Normal | 135 | 63
  NEU Normal, Month 7, Below: number analyzed (Participants) | 152 | 72
  NEU Normal, Month 7, Below | 14 | 8
  NEU Normal, Month 7, Above: number analyzed (Participants) | 152 | 72
  NEU Normal, Month 7, Above | 3 | 1
  NEU Below, Month 2, Normal: number analyzed (Participants) | 13 | 8
  NEU Below, Month 2, Normal | 10 | 5
  NEU Below, Month 2, Below: number analyzed (Participants) | 13 | 8
  NEU Below, Month 2, Below | 3 | 3
  NEU Below, Month 2, Above: number analyzed (Participants) | 13 | 8
  NEU Below, Month 2, Above | 0 | 0
  NEU Below, Month 7, Normal: number analyzed (Participants) | 12 | 8
  NEU Below, Month 7, Normal | 8 | 6
  NEU Below, Month 7, Below: number analyzed (Participants) | 12 | 8
  NEU Below, Month 7, Below | 3 | 2
  NEU Below, Month 7, Above: number analyzed (Participants) | 12 | 8
  NEU Below, Month 7, Above | 1 | 0
  PLA Normal, Month 2, Normal: number analyzed (Participants) | 164 | 78
  PLA Normal, Month 2, Normal | 158 | 68
  PLA Normal, Month 2, Below: number analyzed (Participants) | 164 | 78
  PLA Normal, Month 2, Below | 3 | 2
  PLA Normal, Month 2, Above: number analyzed (Participants) | 164 | 78
  PLA Normal, Month 2, Above | 3 | 2
  PLA Normal, Month 2, Missing: number analyzed (Participants) | 164 | 78
  PLA Normal, Month 2, Missing | 0 | 6
  PLA Normal, Month 7, Normal: number analyzed (Participants) | 163 | 76
  PLA Normal, Month 7, Normal | 156 | 71
  PLA Normal, Month 7, Below: number analyzed (Participants) | 163 | 76
  PLA Normal, Month 7, Below | 2 | 1
  PLA Normal, Month 7, Above: number analyzed (Participants) | 163 | 76
  PLA Normal, Month 7, Above | 5 | 4
  PLA Below, Month 2, Normal: number analyzed (Participants) | 2 | 3
  PLA Below, Month 2, Normal | 0 | 2
  PLA Below, Month 2, Below: number analyzed (Participants) | 2 | 3
  PLA Below, Month 2, Below | 2 | 1
  PLA Below, Month 2, Above: number analyzed (Participants) | 2 | 3
  PLA Below, Month 2, Above | 0 | 0
  PLA Below, Month 7, Normal: number analyzed (Participants) | 2 | 3
  PLA Below, Month 7, Normal | 1 | 0
  PLA Below, Month 7, Below: number analyzed (Participants) | 2 | 3
  PLA Below, Month 7, Below | 1 | 2
  PLA Below, Month 7, Above: number analyzed (Participants) | 2 | 3
  PLA Below, Month 7, Above | 0 | 0
  PLA Below, Month 7, Missing: number analyzed (Participants) | 2 | 3
  PLA Below, Month 7, Missing | 0 | 1
  PLA Above, Month 2, Normal: number analyzed (Participants) | 3 | 3
  PLA Above, Month 2, Normal | 2 | 1
  PLA Above, Month 2, Below: number analyzed (Participants) | 3 | 3
  PLA Above, Month 2, Below | 0 | 0
  PLA Above, Month 2, Above: number analyzed (Participants) | 3 | 3
  PLA Above, Month 2, Above | 1 | 2
  PLA Above, Month 7, Normal: number analyzed (Participants) | 3 | 3
  PLA Above, Month 7, Normal | 0 | 0
  PLA Above, Month 7, Below: number analyzed (Participants) | 3 | 3
  PLA Above, Month 7, Below | 0 | 0
  PLA Above, Month 7, Above: number analyzed (Participants) | 3 | 3
  PLA Above, Month 7, Above | 3 | 3
  RBC Normal, Month 2, Normal: number analyzed (Participants) | 154 | 82
  RBC Normal, Month 2, Normal | 149 | 75
  RBC Normal, Month 2, Below: number analyzed (Participants) | 154 | 82
  RBC Normal, Month 2, Below | 0 | 0
  RBC Normal, Month 2, Above: number analyzed (Participants) | 154 | 82
  RBC Normal, Month 2, Above | 5 | 2
  RBC Normal, Month 2, Missing: number analyzed (Participants) | 154 | 82
  RBC Normal, Month 2, Missing | 0 | 5
  RBC Normal, Month 7, Normal: number analyzed (Participants) | 153 | 80
  RBC Normal, Month 7, Normal | 148 | 78
  RBC Normal, Month 7, Below: number analyzed (Participants) | 153 | 80
  RBC Normal, Month 7, Below | 2 | 1
  RBC Normal, Month 7, Above: number analyzed (Participants) | 153 | 80
  RBC Normal, Month 7, Above | 3 | 1
  RBC Below, Month 2, Normal: number analyzed (Participants) | 2 | 0
  RBC Below, Month 2, Normal | 2 | 0
  RBC Below, Month 2, Below: number analyzed (Participants) | 2 | 0
  RBC Below, Month 2, Below | 0 | 0
  RBC Below, Month 2, Above: number analyzed (Participants) | 2 | 0
  RBC Below, Month 2, Above | 0 | 0
  RBC Below, Month 7, Normal: number analyzed (Participants) | 2 | 0
  RBC Below, Month 7, Normal | 2 | 0
  RBC Below, Month 7, Below: number analyzed (Participants) | 2 | 0
  RBC Below, Month 7, Below | 0 | 0
  RBC Below, Month 7, Above: number analyzed (Participants) | 2 | 0
  RBC Below, Month 7, Above | 0 | 0
  RBC Above, Month 2, Normal: number analyzed (Participants) | 13 | 2
  RBC Above, Month 2, Normal | 7 | 0
  RBC Above, Month 2, Below: number analyzed (Participants) | 13 | 2
  RBC Above, Month 2, Below | 0 | 0
  RBC Above, Month 2, Above: number analyzed (Participants) | 13 | 2
  RBC Above, Month 2, Above | 6 | 1
  RBC Above, Month 2, Missing: number analyzed (Participants) | 13 | 2
  RBC Above, Month 2, Missing | 0 | 1
  RBC Above, Month 7, Normal: number analyzed (Participants) | 13 | 2
  RBC Above, Month 7, Normal | 7 | 0
  RBC Above, Month 7, Below: number analyzed (Participants) | 13 | 2
  RBC Above, Month 7, Below | 0 | 0
  RBC Above, Month 7, Above: number analyzed (Participants) | 13 | 2
  RBC Above, Month 7, Above | 6 | 1
  RBC Above, Month 7, Missing: number analyzed (Participants) | 13 | 2
  RBC Above, Month 7, Missing | 0 | 1
  WBC Normal, Month 2, Normal: number analyzed (Participants) | 155 | 75
  WBC Normal, Month 2, Normal | 142 | 62
  WBC Normal, Month 2, Below: number analyzed (Participants) | 155 | 75
  WBC Normal, Month 2, Below | 7 | 3
  WBC Normal, Month 2, Above: number analyzed (Participants) | 155 | 75
  WBC Normal, Month 2, Above | 6 | 4
  WBC Normal, Month 2, Missing: number analyzed (Participants) | 155 | 75
  WBC Normal, Month 2, Missing | 0 | 6
  WBC Normal, Month 7, Normal: number analyzed (Participants) | 154 | 73
  WBC Normal, Month 7, Normal | 133 | 66
  WBC Normal, Month 7, Below: number analyzed (Participants) | 154 | 73
  WBC Normal, Month 7, Below | 4 | 2
  WBC Normal, Month 7, Above: number analyzed (Participants) | 154 | 73
  WBC Normal, Month 7, Above | 17 | 4
  WBC Normal, Month 7, Missing: number analyzed (Participants) | 154 | 73
  WBC Normal, Month 7, Missing | 0 | 1
  WBC Below, Month 2, Normal: number analyzed (Participants) | 4 | 2
  WBC Below, Month 2, Normal | 4 | 1
  WBC Below, Month 2, Below: number analyzed (Participants) | 4 | 2
  WBC Below, Month 2, Below | 0 | 1
  WBC Below, Month 2, Above: number analyzed (Participants) | 4 | 2
  WBC Below, Month 2, Above | 0 | 0
  WBC Below, Month 7, Normal: number analyzed (Participants) | 4 | 2
  WBC Below, Month 7, Normal | 4 | 2
  WBC Below, Month 7, Below: number analyzed (Participants) | 4 | 2
  WBC Below, Month 7, Below | 0 | 0
  WBC Below, Month 7, Above: number analyzed (Participants) | 4 | 2
  WBC Below, Month 7, Above | 0 | 0
  WBC Above, Month 2, Normal: number analyzed (Participants) | 10 | 7
  WBC Above, Month 2, Normal | 10 | 7
  WBC Above, Month 2, Below: number analyzed (Participants) | 10 | 7
  WBC Above, Month 2, Below | 0 | 0
  WBC Above, Month 2, Above: number analyzed (Participants) | 10 | 7
  WBC Above, Month 2, Above | 0 | 0
  WBC Above, Month 7, Normal: number analyzed (Participants) | 10 | 7
  WBC Above, Month 7, Normal | 9 | 6
  WBC Above, Month 7, Below: number analyzed (Participants) | 10 | 7
  WBC Above, Month 7, Below | 0 | 0
  WBC Above, Month 7, Above: number analyzed (Participants) | 10 | 7
  WBC Above, Month 7, Above | 1 | 1

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days0-6) post-vaccination period. Unsolicited adverse events (AEs): during the 30-day (Days 0-29) post-vaccination period. Serious adverse events (SAEs): Throughout the entire study period (active phase and extended safety follow-up): up to Month 12.
Arm/Group | Cervarix Group | Engerix-B Group
All-Cause Mortality (participants affected / at risk) | 0/181 | 0/89
Serious Adverse Events (participants affected / at risk) | 3/181 | 1/89
Other Adverse Events (participants affected / at risk) | 170/181 | 73/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cervarix Group (N=181) | Engerix-B Group (N=89)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0/175 (0) | 1/86 (1) — This serious adverse event was recorded during the ESFU phase, which only included subjects that could have been contacted by telephone for the Safety follow-up at Month 12, hence the number of participants at risk is different.
Appendicitis (Infections and infestations) | 1/175 (1) | 0/86 (0) — This serious adverse event was recorded during the ESFU phase, which only included subjects that could have been contacted by telephone for the Safety follow-up at Month 12, hence the number of participants at risk is different.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervarix Group (N=181) | Engerix-B Group (N=89)
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 (38) | 10 (13)
Erythema (Skin and subcutaneous tissue disorders) | 51 (87) | 15 (29)
Fatigue (General disorders) | 82 (130) | 42 (61)
Gastrointestinal disorder (Gastrointestinal disorders) | 40 (61) | 14 (19)
Headache (Nervous system disorders) | 82 (131) | 40 (56)
Myalgia (Musculoskeletal and connective tissue disorders) | 88 (142) | 23 (32)
Nasopharyngitis (Infections and infestations) | 12 (13) | 3 (3)
Pain (General disorders) | 159 (378) | 39 (57)
Pyrexia (General disorders) | 39 (56) | 19 (24)
Rash (Skin and subcutaneous tissue disorders) | 16 (20) | 5 (5)
Swelling (General disorders) | 36 (56) | 7 (8)

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.